CLINICAL TRIAL: NCT07245680
Title: Comparison of Initial Dual Oral COMbination Therapy to MOnotherapy in Pulmonary Arterial Hypertension With Cardiovascular comorbiDITIES
Brief Title: COMMODITIES Trial: Initial Dual Oral Therapy vs Monotherapy in PAH With Cardiovascular Comorbidities
Acronym: COMMODITIES
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP230847; 2023-509891-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Comorbidities; Cardiovascular Disease (CVD)
Keywords: PAH; Endothelin Receptor Antagonist (Ambrisentan); Phosphodiesterase-5 Inhibitor (Tadalafil); Cardiovascular Comorbidities; Combination Therapy; Randomized Controlled Trial; Pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Cardiovascular Diseases | interventions — Tadalafil; ambrisentan

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either tadalafil plus ambrisentan or tadalafil plus placebo, in a parallel assignment design with two treatment arms under double-blind masking.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind design: participants and investigators are blinded to treatment allocation. A matching placebo is used in place of ambrisentan to ensure blinding, while tadalafil is given in both arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tadalafil + Ambrisentan (Experimental): Tadalafil - 20 mg once daily for 7 days, then 40 mg once daily (2 × 20 mg tablets). Dose may be reduced to 20 mg once daily if not tolerated.
  Ambrisentan - 5 mg once daily for 4 weeks, then 10 mg once daily (2 × 5 mg tablets). Dose may be maintained at 5 mg once daily in case of intolerance
  Interventions: Drug: Tadalafil; Drug: Ambrisentan
- Tadalafil + Placebo (Active Comparator): Tadalafil - 20 mg once daily for 7 days, then 40 mg once daily (2 × 20 mg tablets). Dose may be reduced to 20 mg once daily if not tolerated.
  Placebo - Matching placebo for ambrisentan, 2 tablets once daily.
  Interventions: Drug: Tadalafil; Drug: Placebo (Ambrisentan-matching)

INTERVENTIONS:
Drug: Tadalafil — Oral phosphodiesterase-5 inhibitor. Initiated at 20 mg once daily for 7 days, then increased to 40 mg once daily (2 × 20 mg tablets). Dose may be reduced to 20 mg once daily if not tolerated.
Drug: Ambrisentan — Oral endothelin receptor antagonist. Initiated at 5 mg once daily for 4 weeks, then increased to 10 mg once daily (2 × 5 mg tablets). Dose may be maintained at 5 mg once daily in case of intolerance.
  Arms: Tadalafil + Ambrisentan
Drug: Placebo (Ambrisentan-matching) — Matching placebo for ambrisentan, 2 tablets once daily, identical in appearance to active drug.
  Arms: Tadalafil + Placebo

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare, progressive disease associated with poor prognosis, especially in patients with cardiovascular comorbidities. Current guidelines recommend initial combination therapy, but evidence is lacking for patients with significant comorbidities who are often excluded from clinical trials.

The COMMODITIES trial is a multicenter, randomized, controlled study designed to compare the efficacy and safety of initial dual oral combination therapy (tadalafil and ambrisentan) versus oral monotherapy in newly diagnosed PAH patients with at least two cardiovascular comorbidities. The study aims to provide robust evidence to guide treatment strategies in this high-risk population.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is characterized by increased pulmonary vascular resistance leading to right heart failure and premature death. Although initial combination therapy with phosphodiesterase-5 inhibitors and endothelin receptor antagonists has demonstrated improved outcomes in patients without major comorbidities, little is known about its benefit-risk balance in patients with cardiovascular comorbidities.

The COMMODITIES study is an investigator-initiated, prospective, randomized, controlled, open-label, phase IV trial conducted under European Regulation (EU) 536/2014. The trial will enroll newly diagnosed PAH patients (confirmed by right heart catheterization) who present with at least two cardiovascular comorbidities (including systemic hypertension, diabetes mellitus, coronary artery disease, obesity, or atrial fibrillation).

Eligible patients will be randomized 1:1 to receive either:

Experimental arm : tadalafil + ambrisentan,

Control arm : : tadalafil +placebo.

The primary endpoint will be the proportion of patients with PAH and cardiovascular comorbidities who achieve after 6 months a low- or an intermediate-low risk profile according to the noninvasive 4-risk strata method as proposed by the 2022 European pulmonary hypertension guidelines.

The total planned sample size is 186, with a study duration of 37 months . Results will provide crucial evidence to inform guideline recommendations and optimize therapeutic strategies in PAH patients with comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Initial PAH diagnosis < 6 months preceding randomisation

  * Negative vasoreactivity test
  * Treatment-naïve PAH (group 1): idiopathic, heritable, associated with drugs and toxin, associated with connective tissue disease, HIV infection or systemic-to-pulmonary congenital shunt corrected for more than one year
  * Meet all of the following hemodynamic criteria by means of a RHC prior to screening:
* mPAP≥25 mmHg and
* PAWP<15 mmHg and
* with PVR≥3 WU

  • Presence of at least two of the following criteria, as listed in the European pulmonary hypertension guidelines:
* History of essential hypertension
* Diabetes mellitus (any type)
* Obesity (defined by a BMI ≥30 kg/m2)
* Coronary heart disease (established by any of the following: history of myocardial infarction, history of percutaneous coronary intervention, angiographic evidence of coronary artery disease (>50% stenosis in ≥1 vessel), positive ST, previous coronary artery bypass graft, stable angina)

  * Participant able to understand the study procedures
  * For women of childbearing potential (WOCBP), effective form of contraception* from screening up to 1 month following discontinuation of the last study treatment
  * Affiliation to the french social security regime
  * Signed written informed consent

Exclusion Criteria:

* Porto-pulmonary hypertension
* Uncorrected systemic-to-pulmonary congenital shunt
* Evidence of thromboembolic disease assessed by ventilation perfusion (V/Q) lung scan or CT pulmonary angiography
* Patients listed for lung or heart-lung transplantation at time of screening
* Patients on any PAH-specific drug therapy at any time preceding randomisation
* Known moderate-to-severe restrictive lung disease (i.e., total lung capacity < 60% of predicted value) or obstructive lung disease (i.e., forced expiratory volume in one second [FEV1] < 60% of predicted, with FEV1 / forced vital capacity < 65%) or known significant chronic lung disease diagnosed by chest imaging (e.g., interstitial lung disease, emphysema).
* Known or suspected pulmonary veno-occlusive disease (PVOD)
* Severe renal insufficiency (creatinine clearance < 30 mL/min)
* Documented severe hepatic impairment (with or without cirrhosis) according to National Cancer Institute organ dysfunction working group criteria, defined as total bilirubin > 3 x ULN or serum AST and/or ALT > 3xULN (assessed by local laboratory at screening) and/or Child-Pugh Class C.
* Haemoglobin < 10 g/dL
* Patient under guardianship curatorship, deprived of liberty
* Pregnant women, or breast-feeding women
* Treatment with other PDE-5i for erectile dysfunction
* Ongoing or planned treatment with nitrates and/or doxazosin.
* Ongoing or planned treatment with riociguat
* Treatment with strong inducers of CYP3A4 (e.g., carbamazepine, rifampin, rifampicin, rifabutin, rifapentin, phenobarbital, phenytoin, and St. John's wort) ≤28 days preceding randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-02-14 (Estimated); Study Completion 2029-02-14 (Estimated)

PRIMARY OUTCOMES:
Mesurement of the risk profile according to the non-invasive 4-risk strata method | Week 24
  Proportion of patients with PAH and with at least two cardiovascular comorbidities who achieve after 24 week a low- or an intermediate-low risk profile according to the non-invasive 4-risk strata method as proposed by the 2022 european pulmonary hypertension guidelines.

SECONDARY OUTCOMES:
Pulmonary vascular resistance | week 24
  Change from baseline to Week 24 in pulmonary vascular resistance, assessed by right heart catheterization and expressed in Wood units (WU).
BNP or NT-proBNP | Week 24
  Percent change from baseline to week 24 in BNP or NT-proBNP
6-Minute Walk Distance (6-MWD) | Week 24
  Change from baseline to week 24 in 6-MWD
WHO/NYHA Functional class | Week 24
  Proportion of participants who improve in WHO/NYHA FC at the end of the DBPC Treatment period
TAPSE/systolic pulmonary artery pressure (SPAP) ratio | Week 24
  Change from baseline to week 24 in the TAPSE/systolic pulmonary artery pressure (SPAP) ratio
Death or Nonfatal Clinical Worsening | Week 24
  Rate of Death or Nonfatal Clinical Worsening defined by hospitalisation for PAH worsening or disease progression defined by worsening of functional class and decrease in 6-min walk distance of more than 15% from baseline, or need for additional specific therapy or lung transplantation
emPHasis-10 score | Week 24
  Change from baseline to week 24 in the emPHasis-10 score
EuroQoL-5 dimensions scale 5 levels (EQ-5D-5L) | Week 24
  Change from baseline to week 24 EuroQoL-5 dimensions scale 5 levels (EQ-5D-5L)
Death | Week 24
  All causes of death

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Bicêtre -Service de pneumologie et soins intensifs respiratoires, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided